CLINICAL TRIAL: NCT00288405
Title: Cordis Neurovascular Feasibility Study of the Enterprise Self-Expanding Stent System to Facilitate Endovascular Coil Embolization of Wide- Neck Saccular Intracranial Artery Aneurysms
Brief Title: The ENTERPRISE Study - Study of the Enterprise Self-Expanding Stent System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Codman & Shurtleff (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN-03-01
Record Dates: First submitted 2005-10-05; First posted 2006-02-08 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-04

CONDITIONS: Aneurysms
Keywords: Intracranial; Wide-neck; Saccular; Aneurysms
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Cordis Self Expanding Stent

SUMMARY:
To evaluate the safety and feasibility of the Cordis Neurovascular Self-Expanding Stent System to facilitate endovascular coil embolization of wide neck saccular intracranial aneurysms.

Cordis Self Expanding Stent for use with embolic coils for the treatment of wide-neck, intracranial, saccular aneurysms arising from a parent vessel

DETAILED DESCRIPTION:
This is a multi-center, prospective, non-randomized feasibility study including 30 subjects. Subjects will receive a safety follow-up evaluation at 30 days (+ two weeks) and an efficacy follow-up evaluation at 6 months (+ four weeks).

ELIGIBILITY:
Inclusion Criteria:

* Patients with intracranial, wide-neck, saccular aneurysms

Exclusion Criteria:

* Subject with Hunt and Hess Grade IV or V subarachnoid hemorrhage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2004-06; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Successful stent placement with satisfactory coil mass position angiographically. | immediately after post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo Boccardi, MD, Principal Investigator — Azienda Ospedaliera
Locations (1):
- Azienda Ospedaliera, Milan, Italy

REFERENCES:
- [Background] Higashida RT, Halbach VV, Dowd CF, Juravsky L, Meagher S. Initial clinical experience with a new self-expanding nitinol stent for the treatment of intracranial cerebral aneurysms: the Cordis Enterprise stent. AJNR Am J Neuroradiol. 2005 Aug;26(7):1751-6. PMID 16091525
- [Result] Weber W, Bendszus M, Kis B, Boulanger T, Solymosi L, Kuhne D. A new self-expanding nitinol stent (Enterprise) for the treatment of wide-necked intracranial aneurysms: initial clinical and angiographic results in 31 aneurysms. Neuroradiology. 2007 Jul;49(7):555-61. doi: 10.1007/s00234-007-0232-2. Epub 2007 May 3. PMID 17476494